CLINICAL TRIAL: NCT04374318
Title: Comparison Study Between Intrathecal and Intravenous Dexmedetomidine in Lower Limb Surgeries
Brief Title: Comparison Between Intrathecal and Intravenous Dexmedetomidine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrhman Alshawadfy, Lecturer of anesthesia and intensive care, Suez Canal University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dex IT IV
Record Dates: First submitted 2020-04-28; First posted 2020-05-05 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Postoperative Analgesia
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IT intrathecal (Active Comparator): administration of intrathecal dexmedetomidine in addition to bupivacaine for lower limb surgeries
  Interventions: Drug: Dexmedetomidine
- IV intravenous (Active Comparator): administration of intravenous dexmedetomidine in addition to spinal anaesthesia for lower limb surgeries
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — INTRATHECAL AND INTRAVENOUS
  Other Names: precidex

SUMMARY:
A prospective, randomized, comparative controlled clinical trial, aiming to compare the use of intrathecal dexmedetomidine by intravenous dexmedetomidine in concern of the first request to analgesia. The secondary end-points were the total postoperative analgesic consumption as well as the VAS.

DETAILED DESCRIPTION:
Seventy patients undergoing lower limb surgeries were included in this study. Using a random number sequence, patients were enrolled in one of two groups: Group T receiving 5 µg of dexmedetomidine (Precedex® 100 µg/mL, Hospira, Inc., IL, U.S.A.) combined with 12.5 mg of 0.5% hyperbaric bupivacaine (Marcaine® Spinal Heavy; Astra, Sodertalje, Sweden) and Group V receiving the same bupivacaine DOSE AND 0.75 microgram/kilogram of body weight dexmedetomidine intravenously. Dexmedetomidine 100 µg/mL was mixed with preservative-free normal saline to 10 µg/mL. The 0.5 mL of dilute dexmedetomidine was added to the bupivacaine in group T. An independent investigator prepared the drug solutions and provided the coded drug to the anaesthetic administrator before the start of the anaesthesia. The anaesthetic administrator, patients, outcome assessors, and data analysts were blinded to the allocation. Spinal Anesthesia Patients were hydrated with 500 mL of 0.9% sodium chloride solution before anaesthesia. The spinal puncture was performed at L3-4 or L4-5 with a midline approach using a 25 G Quincke needle in the lateral decubitus position. After confirmation of free flow and clear cerebrospinal fluid, the drug was administered and the patients were then placed in the supine neutral position.

Assessment: The primary end-point of this study was the first request to analgesia. The secondary end-points were the total postoperative analgesic consumption as well as the VAS.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients
* age 18-65 years
* scheduled for lower limb surgery
* spinal anaesthesia

Exclusion Criteria:

* patients with coagulopathy
* infection at the site of lumbar puncture
* beta-blockers or calcium channel blockers usage
* hypersensitivity to Bupivacaine or Dexmedetomidine
* any other contra-indications for spinal anaesthesia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
First request to analgesia | Postoperative up to 24 hours
  The first time the patient is asking for analgesia to control his pain

SECONDARY OUTCOMES:
Total postoperative analgesia consumption | Postoperative up to 24 hours
  Total consumption of analgesia to control pain
visual analogue scale | Every two hours for 24 hours postoperative
  The score subjectively measures the severity of pain and it is ranging from 0 when there is no pain to 10 when it is the worse pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrhman Alshawadfy, MD, Principal Investigator — Suez Canal University
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No